CLINICAL TRIAL: NCT02870660
Title: Identification of Familial Hypercholesterolemia Amongst Patients With Premature Acute Coronary Syndrome, Follow-up and Treatment
Brief Title: Familial Hypercholesterolemia Amongst Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Isfahan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Golnaz Vaseghi, Research Vice Chancellor, Isfahan University of Medical Sciences
Other Study IDs: IsfahanICRI
Record Dates: First submitted 2016-08-07; First posted 2016-08-17 (Estimated); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: Familial Hypercholesterolemia; Cardiac Event; Acute Coronary Syndrome
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Cardiovascular Diseases; Acute Coronary Syndrome | interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma, buffy coat, blood.

INTERVENTIONS:
Other: Registry

SUMMARY:
Familial hypercholesterolemia (FH) is a most prevalent genetic disorder, defines as high cholesterol level and premature death. The prevalence of FH has been reported in few countries however unknown in Iran. Thus recognize the FH patients, determine the diagnostic strategies and appropriate treatments are important.

Also acute coronary syndrome (ACS) is a group of conditions which arises from reduction of blood flow in coronary arteries. Three specific conditions are included: ST elevation myocardial infarction, non ST elevation myocardial infarction and unstable angina. Premature ACS defined by occurrence of ACS<55 for men and ACS<60 for women. Studies demonstrated direct connection between familial hypercholesterolemia and occurrence of premature ACS. Investigators intent to detection of FH amongst patients with acute coronary syndrome.

DETAILED DESCRIPTION:
Familial hypercholesterolemia (FH) is a genetic disorder, defines as high cholesterol levels, particularly very high levels of low-density lipoprotein (LDL), in the blood and early cardiovascular events and premature death. FH is an autosomal dominant disease with a prevalence of 1:500 (new study in Netherlands demonstrated 1:244) in population more frequent than Cystic fibrosis, mellitus diabetes or neonatal hypothyroidism. Canadian registry demonstrated FH is more common among some specific population such as French Canadian, Christian Lebanese, and Afrikaner descent. The Major causes of FH are pathogenic variant in the LDL-receptor (LDLR) gene or the Apo lipoprotein B (APOB) gene. The clinical signs of FH are high level of Cholesterol (between 350-550 mg/dL in heterozygous), Yellow deposits of cholesterol-rich fat in various places on the body such as around the eyelids (known as xanthelasma palpebrarum), the outer margin of the iris (known as arcus senilis corneae), and in the tendons of the hands, elbows, knees and feet, particularly the Achilles tendon (known as a tendon xanthoma).FH is a hidden syndrome which leads to cardiovascular disease.

Acute coronary syndrome is a term used to describe a range of conditions associated with sudden, reduced blood flow to the heart.

A study in Switzerland has shown that 50% of patients with premature ACS have FH. Thus Investigators can screen FH with high probability amongst patients with acute coronary syndrome.

After introducing the statins total mortality have reduced significantly in these patients. Thus screening and identification of patients and treatment with the most effective therapies will decrease the risk of premature death.

Also, most of patients require an appropriate lipid-lowering medication. Although the genetic problem is the most important factor to expression of FH, other factors like environmental and metabolic factor can be effective in CVD and premature death.

Following scoring of patients, a one-year and 30-day survival model were created in order to assess the effect of elevated cholesterol on survival,.

ELIGIBILITY:
Inclusion Criteria:

* Patients experienced premature cardiac events.

Exclusion Criteria:

* Previously registered FH.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: participating with premature ACS across Isfahan hospitals.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Number of Familial hypercholesterolemia amongst patients with premature acute coronary syndrome. | 1 year

SECONDARY OUTCOMES:
Survival time after hospitalization. | 30 days
Low Density Lipoprotein (LDL-C) at during follow-up. | 1 Year
High Density Lipoprotein (HDL) at during follow-up. | 1 Year
triglycerides (TG) at during follow-up. | 1 Year
LDL-receptor frequency of mutation in Persian Population. | 1 Year
Apo-B frequency of mutation in Persian Population. | 1 Year
PCSK9 frequency of mutation in Persian Population. | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan cardio vascular research instiute, Isfahan, Iran